CLINICAL TRIAL: NCT07094724
Title: High-titer West Nile Virus-neutralizing Plasma for Hospitalized Patients With West Nile Fever: a Prospective Controlled Clinical Study Using Historical Controls
Brief Title: High-Titer Neutralizing Plasma for West Nile Fever in Hospitalized Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gili Regev-Yochay MD (Other Government)
Responsible Party: Sponsor-Investigator, Gili Regev-Yochay MD, Director of the Sheba Pandemic Preparedness Research Institute (SPRI), Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-25-2255-GR-CTIL
Record Dates: First submitted 2025-06-22; First posted 2025-07-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: West Nile Fever
Keywords: West Nile Fever; plasma; neuroinvasive WN disease
MeSH Terms: conditions — West Nile Fever

STUDY DESIGN:
Intervention Model Description: All recruited patients will recieve high neutrlizing plasma, the intervention arm will be compared to historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WN-neutralizing Plasma (Experimental): IV plasma
  Interventions: Biological: Plasma
- historical untreated control (No Intervention)

INTERVENTIONS:
Biological: Plasma — administration of IV high-titer WNV-neutralizing plasma
  Arms: WN-neutralizing Plasma

SUMMARY:
This study will test whether plasma containing high levels of neturalizing antibodies against West Nile virus (WNV) can help people hospitalized with severe West Nile fever recover faster and avoid serious complications. West Nile virus is spread by mosquitoes and can cause mild flu-like symptoms or, in severe cases, brain infections. Currently, there is no specific medication to treat the infection, and doctors primarily provide supportive care.

In this study, patients who are sick enough to require hospitalization will receive plasma donated by people who have recovered from West Nile virus and developed high titer neutralizing antibodies against the disease. Researchers will closely monitor these patients to see how quickly their symptoms improve and whether the plasma helps reduce the risk of death or shorten hospital stays.

To evaluate how well the plasma works, researchers will compare these patients to others who were infected in the past for West Nile virus but did not receive plasma. The study will also examine whether the plasma is safe to use and whether it causes any side effects.

Through this research, scientists hope to determine if antibody-rich plasma could become a helpful treatment option for people with severe West Nile virus infections.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized due to WNF, confirmed by a positive IgM or PCR result in blood or cerebrospinal fluid (CSF).
* Symptomatic acute illness, including fever and/or neurological manifestations (headache, somnolence, confusion, seizures, personality changes, extra-pyramidal manifestations, cranial nerve palsies, etc.).
* No more than 72 hours have elapsed since collection of diagnostic sample.
* Age criteria

  * Age ≥60 years OR
  * Age 18-59 years with previously documented immunosuppression, including hypogammaglobulinemia, treatment with anti-CD20 agents during the last 12 months, hematologic malignancy, bone marrow transplantation, solid organ transplantation, acquired immunodeficiency syndrome (AIDS), or severe primary immunodeficiency.

Exclusion Criteria:

* Age <60 years without significant immunosuppression.
* More than 72 hours have elapsed since collection of diagnostic sample.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within 30 days post enrollment. | 0-30 days

SECONDARY OUTCOMES:
MMSE score at enrollment and at 30 (±3) days post enrollment | 0-33 days
Discharge to pre-hospitalization residence setting. | 0-90 days.
  Patients who were discharged to their pre-hospitalization residence setting will be coded "1"; Patients who were discharged to another setting (e.g., rehabilitation facility) will be coded "0".
Length of hospital stay | 0-90 days.
Serum WNV PCR, IgG, IgM, IgA and neutralizing antibody levels at enrollment, at 7 (±3) days (if still hospitalized), and 30 (±3) days post enrollment. | 0-33 days
WNV PCR, IgG, IgM, IgA and neutralizing antibodies levels in the CSF, at enrollment and within 48-72 (±48) hours post enrollment. | 0-7 days
Serum will be kept for further assessment of additional immunological indices and markers of inflammation. | 10 years.
Peripheral Blood Mononuclear Cell (PBMC) collection at enrollment, at 14 (±3) days (if still hospitalized), and at 30 (±3) days post enrollment. | 0-33 days
Change in Barthel Index at 30 (±3) days post enrollment, compared to baseline. | 0-33 days.
Change in GCS score at 30 (±3) days post enrollment, compared to enrollment. | 0-33 days.

CONTACTS AND LOCATIONS:
Overall Officials: Gili Regev-Yochay, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be available by a reasonable request to the PI, after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: PI & CRA

REFERENCES:
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Teasdale G, Maas A, Lecky F, Manley G, Stocchetti N, Murray G. The Glasgow Coma Scale at 40 years: standing the test of time. Lancet Neurol. 2014 Aug;13(8):844-54. doi: 10.1016/S1474-4422(14)70120-6. PMID 25030516
- [Background] Wade DT, Collin C. The Barthel ADL Index: a standard measure of physical disability? Int Disabil Stud. 1988;10(2):64-7. doi: 10.3109/09638288809164105. PMID 3042746
- [Background] Norris D, Clark MS, Shipley S. The Mental Status Examination. Am Fam Physician. 2016 Oct 15;94(8):635-641. PMID 27929229
- [Background] Katzenellenbogen G, Canetti M, Margalit I, Shusterman Y, Simchovitz-Gesher A, Naveh L, Baharav N, Goldenfeld M, Belkin A, Brod M, Wieder-Finesod A, Leshem E, Magiel E, Levy I, Lustig Y, Indenbaum V, Maggio N, Dekel S, Mechnik B, Peretz Y, Barda N, Tafesh A, Yahav D, Regev-Yochay G. West Nile Virus Outbreak in Israel 2024 Compared with Previous Seasons: A Retrospective Study. Infect Dis Ther. 2025 Jul;14(7):1405-1415. doi: 10.1007/s40121-025-01140-3. Epub 2025 Apr 3. PMID 40180788
- [Background] Popescu CP, Florescu SA, Hasbun R, Harxhi A, Evendar R, Kahraman H, Neuberger A, Codreanu D, Zaharia MF, Tosun S, Ceausu E, Ruta SM, Dragovac G, Pshenichnaya N, Gopatsa G, Shmaylenko O, Nagy E, Malbasa JD, Strbac M, Pandak N, Pullukcu H, Lakatos B, Cag Y, Cascio A, Coledan I, Oncu S, Erdem H. Prediction of unfavorable outcomes in West Nile virus neuroinvasive infection - Result of a multinational ID-IRI study. J Clin Virol. 2020 Jan;122:104213. doi: 10.1016/j.jcv.2019.104213. Epub 2019 Nov 11. PMID 31778945
- [Background] Roberts JA, Kim CY, Hwang SA, Hassan A, Covington E, Heydari K, Lyerly M, Sejvar JJ, Hasbun R, Prasad M, Thakur KT. Clinical, Prognostic, and Longitudinal Functional and Neuropsychological Features of West Nile Virus Neuroinvasive Disease in the United States: A Systematic Review and Meta-Analysis. Ann Neurol. 2025 Jul;98(1):93-106. doi: 10.1002/ana.27220. Epub 2025 Feb 26. PMID 40008684
- [Background] Chancey C, Grinev A, Volkova E, Rios M. The global ecology and epidemiology of West Nile virus. Biomed Res Int. 2015;2015:376230. doi: 10.1155/2015/376230. Epub 2015 Mar 19. PMID 25866777
- [Background] Moirano G, Fletcher C, Semenza JC, Lowe R. Short-term effect of temperature and precipitation on the incidence of West Nile Neuroinvasive Disease in Europe: a multi-country case-crossover analysis. Lancet Reg Health Eur. 2024 Dec 4;48:101149. doi: 10.1016/j.lanepe.2024.101149. eCollection 2025 Jan. PMID 39717226
- [Background] Erazo D, Grant L, Ghisbain G, Marini G, Colon-Gonzalez FJ, Wint W, Rizzoli A, Van Bortel W, Vogels CBF, Grubaugh ND, Mengel M, Frieler K, Thiery W, Dellicour S. Contribution of climate change to the spatial expansion of West Nile virus in Europe. Nat Commun. 2024 Feb 8;15(1):1196. doi: 10.1038/s41467-024-45290-3. PMID 38331945